CLINICAL TRIAL: NCT05707572
Title: Manipulation Versus Steroid Injection in the Treatment of Morton's Neuroma
Brief Title: Morton's Neuroma: Manipulation Versus Steroid Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dundee Podiatry Clinic (Other)
Collaborators: Queen Margaret University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PDN001; 129586 (Registry Identifier: Integrated Reasearch Application System)
Record Dates: First submitted 2018-07-24; First posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Morton Neuroma
Keywords: manipulation; plantar digital neuritis; morton's neuroma; nerve entrapment; foot
MeSH Terms: conditions — Morton Neuroma; Nerve Compression Syndromes | interventions — Methylprednisolone; Methylprednisolone Acetate; Lidocaine; Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- steroid injection (Active Comparator): 1 injection of 1mL methylprednisolone [40mg]with 1 mL 2% lignocaine
  Interventions: Drug: methylprednisolone
- manual manipulation (Experimental): weekly manipulations to the metatarsophalangeal joints of the forefoot for 6 weeks
  Interventions: Procedure: manual manipulation

INTERVENTIONS:
Drug: methylprednisolone — a single injection of 1 mL methylprednisolone [40 mg] and 1 mL 2% lignocaine
  Other Names: Depo-Medrone with Lidocaine (40mg + 10mg)/ml
  Arms: steroid injection
Procedure: manual manipulation — The lesser MTPJs of the affected foot will be manually manipulated using a high velocity, low amplitude thrust technique.
  Other Names: adjustment
  Arms: manual manipulation

SUMMARY:
This study compares manipulative therapy to steroid injection in the treatment of Morton's Neuroma.

DETAILED DESCRIPTION:
The aim of this study is to establish whether manipulative therapy is an effective treatment for Morton's neuroma, a nerve entrapment in the foot. Steroid injection is the current gold standard conservative treatment for this condition. Therefore, a subject group shall be compared to a steroid injection intervention group. Outcomes will be compared using visual analogue pain scales -VAS, Foot Function Index questionnaires and algometric pressure threshold testing. An improvement in the manipulation group VAS of 20mm above the injection group shall be considered as the minimum worthwhile change as this has been identified as the minimum clinically important difference in pain between treatment groups in visual analogue pain scales.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of morton's neuroma
* over 18 years of age
* presenting VAS score > 30mm

Exclusion Criteria:

* diabetes,
* rheumatoid arthritis
* fibromyalgia.
* Those currently taking Statins or analgesics
* previous neuroma surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Visual analogue pain scale | pre treatment at each clinic visit and then 3,6,9 and 12 months
  Measuring changes in self reported pain over time. 100mm scale with anchored prompts of "no pain" at 0mm and "worst pain ever" at 100mm

SECONDARY OUTCOMES:
Algometric pressure threshold meter | pre treatment at each clinic visit and then 3,6,9 and 12 months
  Measuring changes in pressure tolerance over time. A meter which reads how much change in pressure a joint can withstand before it registers discomfort

OTHER OUTCOMES:
Foot function index questionnaire | pre treatment at each clinic visit and then 3,6,9 and 12 months
  A questionnaire to establish subjects level of function, pain and mobility changes over time
Manchester Oxford Foot Pain Questionnaire | pre treatment at each clinic visit and then 3,6,9 and 12 months
  Patient reported outcome measurement tool to measure changes in foot pain over time
Short Form 36 pain and disability Questionnaire | pre treatment at each clinic visit and then 3,6,9 and 12 months
  A quality of life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: David G Cashley, BSc(Hons)Pod, Principal Investigator — Queen Margaret University
Locations (1):
- Podiatry Department NHS Lothian, Edinburgh, Lothian, United Kingdom